CLINICAL TRIAL: NCT07224841
Title: Development of a cfDNA 5mC/5hmC-based Epigenetic Biomarker Panel to Identify Determinants of Response In VEGF/EGFR-targeted Therapy for Metastatic Colorectal Cancer
Brief Title: Development of a cfDNA 5mC/5hmC-based Biomarker Panel to Predict Targeted Therapy Efficacy in mCRC
Acronym: EpiDRIVE
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/EpiDRIVE
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: CRC (Colorectal Cancer)
Keywords: mCRC; Target therapy; 5mc/5hmc; 5-hydroxymethylation; Metastatic colorectal cancer; anti-EGFR therapy; anti-VEGF therapy; RAS/BRAF mutation; 5-methylcytosine
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Discovery Cohort - Long PFS Group (Responder): Patients with metastatic colorectal cancer (mCRC) who received EGFR- or VEGF-targeted therapy and achieved a progression-free survival (PFS) ≥ 12 months, classified as clinical responders.
  Pre-treatment plasma cfDNA samples were analyzed by genome-wide 5mC/5hmC sequencing to identify epigenetic determinants associated with durable treatment response.
  Interventions: Diagnostic Test: cfDNA 5mC/5hmC Sequencing (EpiDRIVE Discovery Phase)
- Discovery Cohort - Short PFS Group (Non-Responder): Patients with mCRC who received EGFR- or VEGF-targeted therapy and showed progression-free survival (PFS) < 12 months, classified as non-responders.
  Pre-treatment cfDNA samples were analyzed using genome-wide 5mC/5hmC sequencing and compared with long-PFS responders to identify differential methylation and hydroxymethylation patterns associated with resistance.
  Interventions: Diagnostic Test: cfDNA 5mC/5hmC Sequencing (EpiDRIVE Discovery Phase)
- Training Cohort - Long PFS Group (Responder): Independent mCRC cohort with PFS ≥ 12 months following EGFR- or VEGF-targeted therapy.
  Candidate cfDNA 5mC/5hmC markers identified in the discovery phase were validated using targeted sequencing (EpiDRIVE assay) to construct the predictive epigenetic biomarker panel.
  Interventions: Diagnostic Test: EpiDRIVE Assay (Targeted Sequencing / qPCR Validation)
- Training Cohort - Short PFS Group (Non-Responder): Independent mCRC patients with PFS < 12 months after targeted therapy. Targeted sequencing using the EpiDRIVE assay was conducted to refine and optimize the predictive model by comparing short- vs long-PFS cases.
  Interventions: Diagnostic Test: EpiDRIVE Assay (Targeted Sequencing / qPCR Validation)
- Validation Cohort - Long PFS Group (Responder): Separate validation cohort of mCRC patients achieving PFS ≥ 12 months under EGFR- or VEGF-targeted therapy.
  qPCR-based EpiDRIVE assay was used to confirm predictive accuracy of the cfDNA 5mC/5hmC biomarker panel in identifying durable responders.
  Interventions: Diagnostic Test: EpiDRIVE Assay (Targeted Sequencing / qPCR Validation)
- Validation Cohort - Short PFS Group (Non-Responder): Independent validation cohort of mCRC patients with PFS < 12 months after targeted therapy.
  cfDNA was analyzed using the qPCR-based EpiDRIVE assay to assess model specificity and distinguish non-responders from long-term responders.
  Interventions: Diagnostic Test: EpiDRIVE Assay (Targeted Sequencing / qPCR Validation)

INTERVENTIONS:
Diagnostic Test: cfDNA 5mC/5hmC Sequencing (EpiDRIVE Discovery Phase) — High-throughput genome-wide sequencing of cfDNA methylation (5mC) and hydroxymethylation (5hmC) profiles from pre-treatment plasma samples in the discovery cohort to identify epigenetic determinants of targeted-therapy response (PFS ≥ 12 months vs < 12 months).
  Groups: Discovery Cohort - Long PFS Group (Responder); Discovery Cohort - Short PFS Group (Non-Responder)
Diagnostic Test: EpiDRIVE Assay (Targeted Sequencing / qPCR Validation) — Targeted sequencing or qPCR-based validation of cfDNA 5mC/5hmC markers identified from the discovery phase to develop and validate a predictive biomarker model discriminating patients with long vs short progression-free survival after EGFR-/VEGF-targeted therapy.
  Groups: Training Cohort - Long PFS Group (Responder); Training Cohort - Short PFS Group (Non-Responder); Validation Cohort - Long PFS Group (Responder); Validation Cohort - Short PFS Group (Non-Responder)

SUMMARY:
The EpiDRIVE study aims to identify cfDNA-based epigenetic determinants of response in metastatic colorectal cancer (mCRC) patients treated with EGFR- or VEGF-targeted therapy.

By integrating 5-methylcytosine (5mC) and 5-hydroxymethylcytosine (5hmC) profiling, this study seeks to develop a predictive biomarker panel capable of differentiating responders from non-responders to targeted therapy.

DETAILED DESCRIPTION:
Metastatic colorectal cancer (mCRC) remains one of the leading causes of cancer-related death. Although targeted agents such as anti-EGFR (cetuximab, panitumumab) and anti-VEGF (bevacizumab) therapies have improved survival, treatment response varies widely even among molecularly defined subgroups.

Traditional biomarkers, including RAS/BRAF mutation and tumor sidedness, fail to accurately predict therapeutic efficacy.

Recent studies highlight the potential of cell-free DNA (cfDNA) methylation (5mC) and hydroxymethylation (5hmC) as sensitive, non-invasive indicators of tumor biology and treatment dynamics.

The EpiDRIVE study integrates cfDNA 5mC/5hmC sequencing and targeted validation to discover and verify epigenetic determinants of therapeutic response.

Discovery phase: Whole-genome 5mC/5hmC profiling to identify differentially modified regions between responders and non-responders.

Training phase: Targeted sequencing to establish a predictive cfDNA epigenetic panel (EpiDRIVE panel).

Validation phase: qPCR-based validation of selected markers in an independent cohort to confirm predictive accuracy.

This study aims to provide a non-invasive biomarker framework to predict and monitor efficacy of EGFR- and VEGF-targeted therapies in mCRC, ultimately guiding personalized treatment selection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal adenocarcinoma (mCRC).
* Received EGFR-targeted therapy (cetuximab/panitumumab) or VEGF-targeted therapy (bevacizumab).
* Availability of pre-treatment plasma sample for cfDNA analysis.
* Documented radiologic response evaluation (RECIST 1.1).
* RAS/BRAF mutation status known.

Exclusion Criteria:

* Inadequate cfDNA quality or low cfDNA yield.
* Non-adenocarcinoma histology.
* Concurrent or prior other active malignancy.
* Active inflammatory or autoimmune disease affecting cfDNA methylation profiles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Stage IV colorectal adenocarcinoma who received EGFR-targeted or VEGF-targeted therapy and had available pre-treatment plasma samples for cfDNA analysis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) according to cfDNA 5mC/5hmC biomarker profile | Up to 36 months from therapy initiation
  Progression-free survival (PFS) among patients with metastatic colorectal cancer (mCRC) receiving EGFR- or VEGF-targeted therapy, stratified by cfDNA 5mC/5hmC-based biomarker status.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 60 months from therapy initiation
  Time from initiation of EGFR- or VEGF-targeted therapy to death from any cause. Overall survival will be analyzed in relation to cfDNA 5mC/5hmC biomarker-defined groups (high vs low EpiDRIVE score) to assess whether epigenetic cfDNA profiles are associated with differences in survival outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data

REFERENCES:
- [Background] Xu C, Mannucci A, Esposito F, Oliveres H, Alonso-Orduna V, Yubero A, Fernandez-Martos C, Salud A, Gallego J, Martin-Richard M, Fernandez-Plana J, Guillot M, Aparicio J, Fakih M, Kopetz S, Feliu J, Maurel J, Goel A. An Exosome-Based Liquid Biopsy Predicts Depth of Response and Survival Outcomes to Cetuximab and Panitumumab in Metastatic Colorectal Cancer: The EXONERATE Study. Clin Cancer Res. 2025 Mar 17;31(6):1002-1015. doi: 10.1158/1078-0432.CCR-24-1934. PMID 39820673
- [Background] Koroukian SM, Booker BD, Vu L, Schumacher FR, Rose J, Cooper GS, Selfridge JE, Markt SC. Receipt of Targeted Therapy and Survival Outcomes in Patients With Metastatic Colorectal Cancer. JAMA Netw Open. 2023 Jan 3;6(1):e2250030. doi: 10.1001/jamanetworkopen.2022.50030. PMID 36656585
- [Background] Tirendi S, Marengo B, Domenicotti C, Bassi AM, Almonti V, Vernazza S. Colorectal cancer and therapy response: a focus on the main mechanisms involved. Front Oncol. 2023 Jul 19;13:1208140. doi: 10.3389/fonc.2023.1208140. eCollection 2023. PMID 37538108
- [Background] Xie YH, Chen YX, Fang JY. Comprehensive review of targeted therapy for colorectal cancer. Signal Transduct Target Ther. 2020 Mar 20;5(1):22. doi: 10.1038/s41392-020-0116-z. PMID 32296018
- [Background] Cai Z, Zhang J, He Y, Xia L, Dong X, Chen G, Zhou Y, Hu X, Zhong S, Wang Y, Chen H, Xie D, Liu X, Liu J. Liquid biopsy by combining 5-hydroxymethylcytosine signatures of plasma cell-free DNA and protein biomarkers for diagnosis and prognosis of hepatocellular carcinoma. ESMO Open. 2021 Feb;6(1):100021. doi: 10.1016/j.esmoop.2020.100021. Epub 2021 Jan 25. PMID 33508734
- [Background] Zeng C, Stroup EK, Zhang Z, Chiu BC, Zhang W. Towards precision medicine: advances in 5-hydroxymethylcytosine cancer biomarker discovery in liquid biopsy. Cancer Commun (Lond). 2019 Mar 29;39(1):12. doi: 10.1186/s40880-019-0356-x. PMID 30922396
- [Background] West-Szymanski DC, Zhang Z, Cui XL, Kowitwanich K, Gao L, Deng Z, Dougherty U, Williams C, Merkle S, He C, Zhang W, Bissonnette M. 5-Hydroxymethylated Biomarkers in Cell-Free DNA Predict Occult Colorectal Cancer up to 36 Months Before Diagnosis in the Prostate, Lung, Colorectal, and Ovarian Cancer Screening Trial. JCO Precis Oncol. 2024 Oct;8:e2400277. doi: 10.1200/PO.24.00277. Epub 2024 Oct 11. PMID 39393034
- [Background] West-Szymanski DC, Zhang Z, Cui XL, Kowitwanich K, Gao L, Deng Z, Dougherty U, Williams C, Merkle S, Moore M, He C, Bissonnette M, Zhang W. Machine learning identifies cell-free DNA 5-hydroxymethylation biomarkers that detect occult colorectal cancer in PLCO Screening Trial subjects. bioRxiv [Preprint]. 2024 Feb 26:2024.02.25.581955. doi: 10.1101/2024.02.25.581955. PMID 38464122
- [Background] Siegel RL, Kratzer TB, Giaquinto AN, Sung H, Jemal A. Cancer statistics, 2025. CA Cancer J Clin. 2025 Jan-Feb;75(1):10-45. doi: 10.3322/caac.21871. Epub 2025 Jan 16. PMID 39817679
- [Background] Song D, Zhang Z, Zheng J, Zhang W, Cai J. 5-Hydroxymethylcytosine modifications in circulating cell-free DNA: frontiers of cancer detection, monitoring, and prognostic evaluation. Biomark Res. 2025 Mar 7;13(1):39. doi: 10.1186/s40364-025-00751-9. PMID 40055844
- [Background] Baldassarre G, L de la Serna I, Vallette FM. Death-ision: the link between cellular resilience and cancer resistance to treatments. Mol Cancer. 2025 May 15;24(1):144. doi: 10.1186/s12943-025-02339-1. PMID 40375296
- [Background] Ferrara R, Imbimbo M, Malouf R, Paget-Bailly S, Calais F, Marchal C, Westeel V. Single or combined immune checkpoint inhibitors compared to first-line platinum-based chemotherapy with or without bevacizumab for people with advanced non-small cell lung cancer. Cochrane Database Syst Rev. 2021 Apr 30;4(4):CD013257. doi: 10.1002/14651858.CD013257.pub3. PMID 33930176
- [Background] Guler GD, Ning Y, Coruh C, Mognol GP, Phillips T, Nabiyouni M, Hazen K, Scott A, Volkmuth W, Levy S. Plasma cell-free DNA hydroxymethylation profiling reveals anti-PD-1 treatment response and resistance biology in non-small cell lung cancer. J Immunother Cancer. 2024 Jan 11;12(1):e008028. doi: 10.1136/jitc-2023-008028. PMID 38212123
- [Background] Shao J, Xu Y, Olsen RJ, Kasparian S, Sun K, Mathur S, Zhang J, He C, Chen SH, Bernicker EH, Li Z. 5-Hydroxymethylcytosine in Cell-Free DNA Predicts Immunotherapy Response in Lung Cancer. Cells. 2024 Apr 19;13(8):715. doi: 10.3390/cells13080715. PMID 38667328
- [Background] Li Q, Huang CC, Huang S, Tian Y, Huang J, Bitaraf A, Dong X, Nevalanen MT, Patel M, Wong J, Zhang J, Manley BJ, Park JY, Kohli M, Gore EM, Kilari D, Wang L. 5-hydroxymethylcytosine sequencing in plasma cell-free DNA identifies unique epigenomic features in prostate cancer patients resistant to androgen deprivation therapies. medRxiv [Preprint]. 2024 Oct 17:2023.10.13.23296758. doi: 10.1101/2023.10.13.23296758. PMID 37904926